CLINICAL TRIAL: NCT05896410
Title: Comparison of Using 3D-Printed Hand Orthosis Versus Thermoplastic Orthosis in Patients With Thumb Carpo-metacarpal Osteoarthritis: A Pilot Randomized Trial Cross-over Study
Brief Title: 3D-Printed Hand Orthosis Versus Thermoplastic Orthosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 122173
Record Dates: First submitted 2023-01-25; First posted 2023-06-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Thumb Osteoarthritis; CMC; Splints
Keywords: Thumb osteoarthrities; CMC; Splint; 3D print; low temprature thermoplastic
MeSH Terms: interventions — Splints; Orthotic Devices

STUDY DESIGN:
Intervention Model Description: In this study, participants act as their controls; traditional orthosis and 3D-printed orthoses. The order of intervention and testing conditions will be determined by drawing a concealed envelope from a bag . The testing protocol will be started after the fitting of orthoses. Participants will use the first orthosis for three weeks, be given a week for washout, and then cross over to the second orthosis. The participants should use the second orthosis for three weeks. All participants will be informed about the research details, and the measurements will be explained and demonstrated to the participant and provided signed informed consent before participation. Patients will receive identical orthotic-wearing instructions. Patients will be asked to use the orthosis during the daytime functional activities and ADLs for at least half of their waking hours. All patients will be asked to report any pain, discomfort, or skin irritations when using the orthosis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thermoplastic Splint(orthosis) (Active Comparator): A static hand-based splint (orthosis) made with a thermoplastic material that immobilizes the CMC and MCP joint will be used.
  Interventions: Device: splint (orthosis)
- 3D printed splint (orthosis) (Experimental): A static hand-based 3D-printed splint (orthosis) made with 3D printing that immobilizes both the CMC and MCP joint will be used.
  Interventions: Device: splint (orthosis)

INTERVENTIONS:
Device: splint (orthosis) — 3D printed splint (orthosis) help prevent the joint from shifting during pinch activities. This reduces improper joint loading and helps reduce pain and the progression of degenerative change in patients with OA.
  Other Names: 3D printed splint (orthosis)

SUMMARY:
This study will investigate the effectiveness of 3D-printed splints for treating thumb osteoarthritis (CMC OA). These splints are made by Occupational Therapists and Physical Therapists out of low-temperature plastic and formed on the patient's hand. 3D printed splints involve photographing the hand and creating a digital file of the splint. This is then printed and fit on the patient.

The goal of this cross-over clinical trial is to compare the effectiveness of 3D-printed splints versus thermoplastic splints for treating thumb osteoarthritis (CMC OA).

The main question[s] it aims to answer are:

Primary objective:

• Evaluate the general useability and possible benefits of splint production by 3D printing in a clinical setting

Secondary objectives:

* Compare the effectiveness of 3D printed orthosis and the low-temperature plastic fabrication manual method in pain reduction
* Compare the effectiveness of 3D printed orthosis and the low-temperature plastic fabrication manual method in improving the function.
* Compare the satisfaction of patients with the 3D printed orthosis and low-temperature plastic fabrication manual method.
* Compare the length of time needed to fabricate each orthosis
* Compare the weight of orthosis

Participants will provide with two splints (traditional orthosis and 3D-printed orthoses). Participants will use the first orthosis for three weeks, be given a week for washout, and then cross over to the second orthosis.

DETAILED DESCRIPTION:
Non-surgical treatment is the initial consideration for symptomatic carpometacarpal (CMC) osteoarthritis (OA). Immobilization with orthosis (splint) is one of the methods of non-surgical treatment. The evidence is mounting regarding the effectiveness of orthosis in OA of the thumb. A recent systematic review indicated that splinting causes a moderate to large effect on pain. However, a recent network meta-analysis showed that a short thermoplastic CMC splint is the best treatment to increase function.

The variations of the recommended orthosis for immobilization of the CMC are varied from the neoprene splints to the rigid thermoplastic material. However, the patient's satisfaction with these materials is different. Patients reported more satisfaction with neoprene thumb splints but found custom-made splints more functional.

Hand therapists typically use low-temperature thermoplastic materials (LTTP) for orthosis fabrication.

3D-printed orthoses are emerging as an alternative for immobilizing joints. Different studies tried to compare the two methods of the 3D printed orthosis with a thermoplastic orthosis and reported some advantages for a 3D printed orthosis. These studies reported advantages including being lighter in weight, producing less incidence of skin irritation, offering better hygiene with less odour and perspiration, appealing and custom-tailored aesthetic design, and the ability to use recycled affordable materials. Furthermore, the fabrication of thermoplastic orthosis needs expertise and knowledge, which require specialized training to fabricate and are time-consuming, expensive, difficult to keep clean, bulky, cumbersome, and unable to tolerate moisture at high temperatures. Also, the thermoplastic material is subject to cracking, requiring the patient to go through the healthcare system again and return to the clinic just for a therapist to make another splint. Off-the-shelf splints have better breathability and longevity but cost more and are often less form-fitting or stabilizing than a therapist-made splint. Despite the numerous advantages of the 3D printed splint listed in the literature, the high cost of equipment, lack of training and skill of clinicians and the long time required for production limited their use in hand therapy.

Progress has been made in developing the 3D of orthoses. Potential advantages include comfort, well-fitting, adequate ventilation in the splint and a clean production process. However, there are challenges in reducing the reliance on the in-person evaluation given the complex geometries of the hand, unavailability of high-resolution scanners, fabrication time that may require multiple visits and cost, equipment materials and expertise. Accurate and high-resolution 3D scanners are available on the market and are currently used in research studies. Different scanners are being used in the literature to scan the hand. Different steps are required to fabricate a 3D printed orthosis, including scanning the body segment with a 3D scanner, CT scan or MRI; transferring the scanned data to a computer modelling software program; printing the orthosis; and finishing/adjusting the final product. The time needed to scan the affected upper limb ranged from 1 to 3 minutes. The time needed to modify the scanned digital file in a computer-aided design software program to be ready for 3D printing was reported to take approximately 1 hour. Only one study reported a 53% reduction in total fabrication time with a 3D-printed orthosis compared with a traditional orthosis.

Few studies compared 3D-printed orthosis with traditional orthosis fabrication in the clinical setting. The reported outcome measures are Outcome measures pain, overall satisfaction, and function. More satisfaction, less skin irritation, itchiness and odour; however, none utilize patients with CMC OA as participants. Chu et al. used 3D hand parametric modelling techniques to create customized designs of short thumb orthoses in healthy adults. They reported that the 3D-printed orthosis provided greater flexibility of hand movement and stronger support than the traditional, manually formed orthosis.

There is a gap in evidence regarding the clinical utility and feasibility of using 3D printing versus traditional orthosis in patients with CMC joint OA.

ELIGIBILITY:
Patients would be eligible to participate in our study :

* At least 18 years old,
* able to provide written informed consent
* indicating immobilization of CMC as part of their therapy. The orthosis treatment can be in any part of their treatment (first users or the patients with experience of using orthosis).

Patients will be excluded if

* have skin irritation, blister, or wound.
* have neurologic conditions affecting their pain perception in the upper limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and general useability | At six weeks
  The feasibility of splint production by 3D printing in a clinical setting will be evaluated by evaluating the degree to which a new intervention is considered suitable, satisfying, or with The Quebec User Evaluation of Satisfaction with Assistive Technology 2(QUEST-2) questionnaire. It is a 12-item outcome measure that assesses user satisfaction with two components, Devices and Services. Psychometric properties have been tested with respect to test-retest stability, alternate-form equivalence, internal consistency, factorial composition and nomological validity. Each item of the QUEST is scored on a 5-point satisfaction scale of zero to 5, which the score for fully agreeing being "5". The score ranges from 0-60, with a higher score indicating more satisfaction with Assistive Technology.

SECONDARY OUTCOMES:
Changes in hand Function | baseline and after each orthosis use((three weeks and six weeks))
  The shortened form of the Disability of the Arm, Shoulder, and Hand Questionnaire (Quick DASH) will be used to measure the upper extremity function . This tool consists of 11 items and a total score ranging from 0 to 100, where 0 indicates no limitation and 100 suggests full disability. Eight questions inquire about the patient's ability to perform certain daily activities.
weight of splint (orthosis) | after each orthosis preperation(baseline)
  will be evaluated by Gram
preparation time for each splint | after each orthosis preperation (baseline)
  length of the time will be recorded for each splint (orthosis).
Change of Pain at CMC joint | baseline and after each orthosis use(three weeks and six weeks)
  Pain will be evaluated by the Numeric Rating Scale (NRS).The NRS is a reliable instrument with demonstrated sensitivity to changes in pain in patients with chronic inflammatory or degenerative pain.

IPD SHARING:
Plan to Share IPD: No